CLINICAL TRIAL: NCT03062319
Title: Optimal Antithrombotic Therapy in Ischemic Stroke Patients with Non-Valvular Atrial Fibrillation and Atherothrombosis
Acronym: ATIS-NVAF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated at the planned interim analysis for futility on July 18, 2023.
Sponsor: National Hospital Organization Osaka National Hospital (Other)
Collaborators: Network for Clinical Stroke Trials (Unknown); The BMS/Pfizer Japan Thrombosis Investigator Initiated Research Program (Unknown)
Responsible Party: Principal Investigator, Hiroshi Yamagami, Director, Department of Stroke Neurology, National Hospital Organization Osaka National Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATIS-NVAF
Record Dates: First submitted 2017-02-08; First posted 2017-02-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke; Atrial Fibrillation; Atherothrombosis
Keywords: anticoagulant; antiplatelet
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Thrombosis | interventions — Anticoagulants; Platelet Aggregation Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual-therapy group (Active Comparator): Dual-therapy group: single anticoagulant drug and single antiplatelet drug. The dosage is determined according to each drug's package insert in Japan. In patients treated with warfarin, the target international normalized ratio (INR) range of 2.0-3.0 for those <70 years and 1.6-2.6 for those =>70 years is recommended according to the Japanese guidelines.
  Interventions: Drug: Oral Anticoagulant; Drug: Antiplatelet Drug
- Single-therapy group (Active Comparator): Single-therapy group: single anticoagulant drug. The dosage is determined according to each drug's package insert in Japan. In patients treated with warfarin, the target international normalized ratio (INR) range of 2.0-3.0 for those <70 years and 1.6-2.6 for those =>70 years is recommended according to the Japanese guidelines.
  Interventions: Drug: Oral Anticoagulant

INTERVENTIONS:
Drug: Oral Anticoagulant — warfarin, dabigatran, rivaroxaban, apixaban, or edoxaban
Drug: Antiplatelet Drug — aspirin, clopidogrel, prasugrel, ticlopidine, or cilostazol
  Arms: Dual-therapy group

SUMMARY:
The Purpose of this open-label randomized controlled multicenter trial is to evaluate the efficacy and safety of mono-drug therapy with oral anticoagulant compared to combination therapy with antiplatelet drug, in ischemic stroke patients with non-valvular atrial fibrillation and atherothrombosis.

DETAILED DESCRIPTION:
The Purpose of this open-label randomized controlled multicenter trial is to evaluate the efficacy and safety of mono-drug therapy with oral anticoagulant compared to combination therapy with antiplatelet drug, in ischemic stroke patients with non-valvular atrial fibrillation and atherothrombosis. Target sample size is 400. The primary outcome is a composite endpoint of ischemic cardiovascular events (cardiovascular death, ischemic stroke, myocardial infarction, systemic embolism, ischemic events requiring urgent revascularization) and major bleeding defined by the International Society on Thrombosis and Haemostasis(ISTH) criteria within 2 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an acute ischemic stroke or TIA from 8 days and up to 360 days from the onset of symptoms
2. Age 20 or older
3. Patients with non-valvular atrial fibrillation (chronic or paroxysmal) who start or continue taking an oral anticoagulant
4. Patients who have one of the following atherothrombotic diseases

   1. A past history of ischemic heart disease (myocardial infarction, angina pectoris, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI)
   2. A past history of peripheral artery disease (symptomatic peripheral arterial occlusive disease, lower extremity bypass surgery/angioplasty/stenting)
   3. Carotid artery stenosis (symptomatic or asymptomatic (=>50% diameter), a history of carotid artery stenting (CAS) or carotid endarterectomy (CEA))
   4. Intracranial artery stenosis (=>50% stenosis of the diameter of a major intracranial artery: intracranial internal carotid artery, anterior cerebral artery (ACA)-A1 and A2, middle cerebral artery (MCA)-M1 and M2, posterior cerebral artery (PCA)-P1 and P2, vertebral artery, and basilar artery; a history of intracranial stent placement or intracranial bypass surgery)
   5. A past history of atherothrombotic brain infarction, lacunar infarction, or branch atheromatous disease
5. Patients without severe disability (modified Rankin Scale score =<4)
6. Patients who can take oral medications
7. Patients who can receive follow-up survey
8. Provision of written informed consent either directly or by a suitable surrogate

Exclusion Criteria:

1. History of myocardial infarction or acute coronary syndrome within the past 12 months
2. Patients who underwent PCI with drug-eluting stents within the past 12 months or PCI with bare-metal stents within the past 3 months
3. Patients who underwent carotid artery stent placement, intracranial stent placement, or lower extremity stent placement within the past 3 months
4. History of symptomatic intracranial hemorrhage or gastrointestinal bleeding within the past 6 months
5. Hemorrhagic diathesis or blood coagulation disorders
6. Platelet counts <100,000 /mm3 at enrollment.
7. Severe anemia (hemoglobin <7 g/dL)
8. Severe renal failure (creatinine clearance =<15 mL/min) or undergoing chronic hemodialysis.
9. Severe liver dysfunction (Grade B or C of the Child-Pugh classification)
10. Patients with severe disability requires constant nursing care, bedridden (modified Rankin Scale score =5)
11. Pregnant or possibly pregnant women
12. Active cancer
13. Expectation of survival less than 2 years
14. Anticoagulant or antiplatelet is scheduled to be discontinued for more than 4 weeks during the follow-up period
15. Planned revascularization procedure during the follow-up period
16. Patients who are enrolled in other trials
17. Patients judged as inappropriate for this study by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of ischemic cardiovascular events and major bleeding | 2 years after randomization
  One of the following ischemic cardiovascular events (cardiovascular death, ischemic stroke, myocardial infarction, systemic embolism, or ischemic events requiring urgent revascularization), or major bleeding defined by the International Society on Thrombosis and Haemostasis (ISTH) criteria

SECONDARY OUTCOMES:
All-cause mortality | 2 years after randomization
  All-cause mortality
Ischemic cardiovascular events | 2 years after randomization
  Ischemic cardiovascular events (cardiovascular death, ischemic stroke, myocardial infarction, systemic embolism, ischemic events requiring urgent revascularization)
All ischemic cardiovascular events including transient ischemia | 2 years after randomization
  All ischemic cardiovascular events including transient ischemia (cardiovascular death, ischemic stroke, transient ischemic attack (TIA), myocardial infarction, unstable angina pectoris, systemic embolism, progression of symptomatic peripheral artery disease, ischemic events requiring urgent revascularization)
Ischemic stroke | 2 years after randomization
  Ischemic stroke
Myocardial infarction and cardiovascular death | 2 years after randomization
  Myocardial infarction and cardiovascular death
major bleeding | 2 years after randomization
  major bleeding defined by the International Society on Thrombosis and Haemostasis (ISTH) criteria
Intracranial hemorrhage | 2 years after randomization
  Intracranial hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Yamagami, MD, Principal Investigator — National Hospital Organization Osaka National Hospital
Locations (1):
- National Hospital Organization Osaka National Hospital, Osaka, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Okazaki S, Tanaka K, Yazawa Y, Doijiri R, Koga M, Ihara M, Yamamoto S, Kamiyama K, Honda Y, Uchida K, Yoshimoto T, Asakura K, Omae K, Tanaka K, Maeda H, Yamamoto H, Hirano T, Toyoda K, Iguchi Y, Noguchi T, Okada Y, Kitagawa K, Sakai N, Yamagami H; ATIS-NVAF Trial Investigators. Optimal Antithrombotics for Ischemic Stroke and Concurrent Atrial Fibrillation and Atherosclerosis: A Randomized Clinical Trial. JAMA Neurol. 2025 Dec 1;82(12):1227-1234. doi: 10.1001/jamaneurol.2025.3662. PMID 41051787
- [Derived] Okazaki S, Yamamoto H, Asakura K, Omae K, Maeda H, Tanaka K, Yamamoto S, Hirano T, Iguchi Y, Sakaguchi M, Koga M, Ihara M, Toyoda K, Noguchi T, Sakai N, Yamagami H. Optimal antithrombotic therapy in ischemic stroke patients with non-valvular atrial fibrillation and atherothrombosis: study protocol for a randomized controlled trial. Front Neurol. 2024 Oct 23;15:1468523. doi: 10.3389/fneur.2024.1468523. eCollection 2024. PMID 39539664